CLINICAL TRIAL: NCT06957561
Title: An Open-Label, Single-Arm Phase Ib/II Clinical Trial to Evaluate the Efficacy and Safety of Disitamab Vedotin Combined With Ivonescimab in the Perioperative Treatment of Cisplatin-Ineligible Muscle-Invasive Bladder Cancer (MIBC)
Brief Title: Disitamab Vedotin Combined With Ivonescimab in Cisplatin-Ineligible Muscle-Invasive Bladder Cancer
Acronym: DIVON
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-094-01
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer; Muscle-invasive Bladder Cancer
Keywords: Cisplatin-Ineligible; Muscle-invasive bladder cancer; Disitamab Vedotin; Ivonescimab; Perioperative treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — disitamab vedotin; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin Combined with Ivonescimab (Experimental): Participants will receive Disitamab Vedotin (2.0 mg/kg, every 2 weeks) for 6 cycles, combined with Ivonescimab (20 mg/kg, every 3 weeks) for 4 cycles, with a total duration of 12 weeks for the neoadjuvant treatment phase. Following the completion of neoadjuvant therapy, participants will undergo radical cystectomy with pelvic lymph node dissection 4-6 weeks after the last dose. In the postoperative adjuvant phase, participants will receive Disitamab Vedotin (2.0 mg/kg, every 3 weeks, for 4 cycles) combined with Ivonescimab (20 mg/kg, every 3 weeks, for 9 cycles), starting 4-8 weeks after surgery.
  Interventions: Drug: Disitamab Vedotin Injection; Drug: Ivonescimab（AK112，a PD-1/VEGF bispecific antibody）; Procedure: Radical Cystectomy with Pelvic Lymph Node Dissection

INTERVENTIONS:
Drug: Disitamab Vedotin Injection — Participants will receive Disitamab Vedotin at a dose of 2.0 mg/kg. In the neoadjuvant phase, it will be administered every 2 weeks for 6 cycles (12 weeks total). In the postoperative adjuvant phase, it will be administered every 3 weeks for 4 cycles, starting 4-8 weeks after surgery.
  Other Names: RC48-ADC
Drug: Ivonescimab（AK112，a PD-1/VEGF bispecific antibody） — Participants will receive Ivonescimab at a dose of 20 mg/kg. In the neoadjuvant phase, it will be administered every 3 weeks for 4 cycles (12 weeks total). In the postoperative adjuvant phase, it will be administered every 3 weeks for 9 cycles, starting 4-8 weeks after surgery.
  Other Names: AK112
Procedure: Radical Cystectomy with Pelvic Lymph Node Dissection — Participants will undergo radical cystectomy with pelvic lymph node dissection 4-6 weeks after the last dose of neoadjuvant treatment.

SUMMARY:
This is a single-arm, open-label, Phase Ib/II clinical trial designed to evaluate the efficacy and safety of Disitamab Vedotin combined with Ivonescimab in the perioperative treatment of cisplatin-ineligible patients with muscle-invasive bladder cancer (MIBC). The study will enroll MIBC patients scheduled for radical cystectomy who have not received prior immunotherapy, targeted therapy, or biological therapy, except for cisplatin chemotherapy. The trial will consist of a neoadjuvant treatment phase (Disitamab Vedotin and Ivonescimab), followed by surgery and an adjuvant treatment phase. Primary efficacy endpoints include the pathological complete response (pCR) rate, while secondary endpoints include disease-free survival, recurrence-free survival, overall survival, and clinical objective response rate. Safety will be monitored throughout the study, and biomarker testing (HER2 and PD-L1) will be conducted to assess treatment efficacy. The study aims to explore the potential of this combination therapy in improving outcomes for MIBC patients.

DETAILED DESCRIPTION:
This open-label, single-arm Phase Ib/II clinical trial aims to assess the efficacy and safety of combining Disitamab Vedotin with Ivonescimab for treating muscle-invasive bladder cancer (MIBC) in patients who are ineligible for cisplatin-based chemotherapy. The trial consists of two primary phases: a safety run-in phase and subsequent treatment phases (neoadjuvant and postoperative adjuvant).

Study Phases:

Safety Run-In Phase:

The first 6 participants will receive an initial dose of Disitamab Vedotin (2.0 mg/kg) and Ivonescimab (20 mg/kg). If ≥2 dose-limiting toxicities (DLTs) occur, dose adjustments will be made (Disitamab Vedotin reduced to 1.5 mg/kg, Ivonescimab to 15 mg/kg). If no significant toxicity occurs, the trial will continue with the original doses.

Neoadjuvant Phase:

Participants will receive 6 cycles of Disitamab Vedotin (2.0 mg/kg, Q2W) and 4 cycles of Ivonescimab (20 mg/kg, Q3W) over 12 weeks. After treatment, patients will undergo radical cystectomy with pelvic lymph node dissection.

Postoperative Adjuvant Phase:

Following surgery, patients will receive 4 cycles of Disitamab Vedotin (2.0 mg/kg, Q3W) and 9 cycles of Ivonescimab (20 mg/kg, Q3W) to reduce the risk of recurrence.

Evaluation:

Tumor Response:

Tumor assessments will be conducted using RECIST 1.1 criteria in the neoadjuvant phase, with imaging follow-up every 12 weeks during the adjuvant phase. The primary endpoint is the objective response rate (ORR).

Biomarker Correlation:

HER2 and PD-L1 expression levels will be assessed as secondary objectives to evaluate their correlation with treatment outcomes.

Safety Monitoring and Data Management:

Adverse events will be documented and evaluated. Regular data checks will ensure the integrity and completeness of patient data. A strict confidentiality protocol will be followed, ensuring the protection of participant information.

Study Population:

Approximately 30 patients with MIBC who are ineligible for cisplatin chemotherapy will be enrolled. Inclusion criteria include documented HER2 expression and eligibility for transurethral resection and radical cystectomy.

Statistical Analysis:

Descriptive statistics will summarize baseline characteristics and treatment outcomes. Kaplan-Meier methods will be used to analyze progression-free survival (PFS) and overall survival (OS), while regression analysis will assess biomarker correlations.

Conclusion:

This trial will provide valuable insights into the potential of Disitamab Vedotin and Ivonescimab as a perioperative treatment for cisplatin-ineligible MIBC patients, offering a new therapeutic option for this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign an informed consent form.
2. Male or female, aged ≥18 years.
3. Expected survival ≥12 weeks.
4. Pathologically confirmed muscle-invasive bladder urothelial carcinoma (MIBC), with the primary pathological component being urothelial carcinoma ≥50%, and no upper urinary tract urothelial carcinoma.
5. Clinical staging (cT2-T4a, N0-1, M0) with no distant metastasis as evaluated by imaging.
6. Based on urologist's assessment, the subject is able to tolerate transurethral resection and radical cystectomy.
7. No prior immunotherapy, targeted therapy, or biological therapy for MIBC. Cisplatin-ineligible patients may be enrolled.
8. Cisplatin chemotherapy intolerance/non-eligibility (defined as CrCl <60 mL/min, ≥2-grade hearing impairment, ≥2-grade peripheral neuropathy, ECOG performance status of 2).
9. Investigator-confirmed HER2 expression: IHC 1+, 2+, or 3+.
10. ECOG performance status 0-2.
11. Adequate cardiac, bone marrow, liver, and renal function, with the following parameters meeting the criteria within 7 days prior to the first dose of study drug (normal values based on the clinical trial center):

    * Left ventricular ejection fraction ≥50%;
    * Hemoglobin ≥9 g/dL;
    * Absolute neutrophil count (ANC) ≥1.5 × 10^9/L;
    * Platelet count ≥90 × 10^9/L;
    * Total bilirubin ≤1.5 times the upper limit of normal (ULN);
    * ALT and AST ≤2.5 × ULN (ALT, AST ≤5 × ULN for patients with liver metastasis);
    * Serum creatinine ≤2.0 × ULN or estimated creatinine clearance (CrCl) ≥30 mL/min based on the Cockcroft-Gault formula;
    * Urine protein <2+ or 24-hour urine protein <1.0g;
    * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5 × ULN.
12. Female subjects must be surgically sterile, postmenopausal, or agree to use at least one medically accepted form of contraception during the study and for 6 months after the treatment period (e.g., intrauterine device, birth control pills, or condoms). A negative pregnancy test must be confirmed within 7 days prior to study enrollment, and subjects must not be breastfeeding. Male subjects must agree to use at least one medically accepted form of contraception during the study and for 6 months after the treatment period.
13. Willing and able to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Prior systemic antitumor treatment, other than cisplatin, such as targeted therapy, immunotherapy, or biological therapy, before the start of study medication.
2. Major surgery within 4 weeks prior to the start of study medication.
3. Positive serum virology tests (based on normal values of the study center):

   * HBsAg or HBcAb positive, with positive HBV DNA copy number.
   * Positive HCVAb (only if HCV RNA PCR test is negative, the subject may be eligible).
   * Positive HIVAb.
4. Receipt of live vaccines within 4 weeks prior to the start of study medication or plans to receive any vaccines during the study (except for the COVID-19 vaccine).
5. Heart failure classified as NYHA class 3 or higher.
6. Known central nervous system metastases.
7. Serious arterial or venous thrombosis, or cardiovascular events such as deep vein thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc., within 1 year before the study medication. Excluding asymptomatic lacunar infarctions that do not require clinical intervention.
8. Active or progressive infections requiring systemic treatment, such as active tuberculosis.
9. Systemic diseases that are not well controlled, as determined by the investigator, including diabetes, hypertension, liver cirrhosis, interstitial lung disease, obstructive lung disease, etc.
10. History of serious bleeding disorders or coagulation abnormalities.
11. History of gastrointestinal perforation or fistula related to anti-VEGF therapy; gastrointestinal perforation, fistula, or intra-abdominal abscess within 3 months before the first dose.
12. History of esophageal or gastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, fistulas, bowel obstruction, intra-abdominal abscess, acute gastrointestinal bleeding, extensive bowel resection (partial colon resection or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea within 6 months before the first dose.
13. Non-healing or poorly healing wounds, active ulcers.
14. Imaging or clinical evidence of current gastrointestinal obstruction, including partial obstruction.
15. Incomplete resolution of prior antitumor treatment toxicity, defined as failure to return to NCI CTCAE v5.0 Grade 0 or 1 toxicity.
16. Active autoimmune disease requiring systemic treatment (e.g., immunosuppressive agents, corticosteroids, or immunomodulators) prior to the start of study medication. The use of related replacement therapy (e.g., thyroid hormone, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
17. History of any other malignant tumors within the past 5 years, except for the following:

    * Malignant tumors expected to be cured after treatment (including but not limited to fully treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery).
18. History of allogeneic hematopoietic stem cell transplant or organ transplant.
19. Prior treatment with PD-(L)1 inhibitors or other antibody-drug conjugates.
20. Known allergies to recombinant humanized anti-HER2 monoclonal antibody MMAE conjugates, PD-1/L1 monoclonal antibodies, VEGF antibodies, other monoclonal antibodies, or their components.
21. Pregnant or breastfeeding women.
22. Any other disease, metabolic abnormalities, abnormal physical examination, or laboratory findings that, in the investigator's judgment, may indicate a condition that is not suitable for study drug use or may affect the interpretation of study results, or place the patient at high risk.
23. Estimated non-compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | 4 months
  The percentage of patients who achieve a pathological complete response (pT0N0) after surgery following neoadjuvant treatment with Disitamab Vedotin combined with Ivonescimab.

SECONDARY OUTCOMES:
Pathological Response Rate | 4 months
  The percentage of patients with pathological complete response (pT0N0) or pathological partial response (≤ ypT1N0M0) during surgery.
1-3 Year Disease-Free Survival (DFS) Rate | Up to 3 years
  The percentage of patients who remain free from local or distant recurrence, or death from any cause, as confirmed by imaging or pathological examination, at 1, 2, or 3 years after surgery.
Recurrence-Free Survival (RFS) | Up to first recurrence of disease or up to 5 years
  The rate of recurrence of the disease after completion of treatment as confirmed by imaging or clinical evidence.
Overall Survival (OS) | Up to death or up to 5 years
  The time from the first dose of neoadjuvant treatment to death from any cause.
Clinical Objective Response Rate (ORR) | Up to 5 years
  Tumor evaluations will be conducted according to RECIST 1.1 criteria for all patients with evaluable lesions at baseline, and responses will be assessed at each tumor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuowei Liu, M.D Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No